CLINICAL TRIAL: NCT01383733
Title: A Phase I Multiple Ascending Dose (MAD) Study of RO5458640, a Humanized Monoclonal Antibody Against the TNF-like Weak Inducer of Apoptosis (TWEAK) Ligand, in Patients With Advanced Solid Tumors
Brief Title: A Study of RO5458640 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP25448
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: RO5458640

INTERVENTIONS:
Drug: RO5458640 — Multiple ascending doses intravenously, weekly or every 2 weeks or every 3 weeks

SUMMARY:
This multicenter, open-label, multiple ascending dose study will evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of RO5458640 in patients with advanced solid tumors. Cohorts of patients will receive ascending doses of RO5458640 intravenously, either weekly or every 2 weeks or every 3 weeks, until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically confirmed malignant solid tumors
* Measurable and/or evaluable disease according to RECIST 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Prior chemotherapy, radiotherapy, or hormonal therapy for cancer within 3 weeks of first study treatment, except for short course palliative radiotherapy for pain
* Antibody therapy or other immunotherapy currently or less than 21 days prior to study treatment
* Current immunosuppressive therapy, including those prescribed for organ transplantation and rheumatologic disease
* Corticoid therapy > 10 mg/day prednisone or equivalent
* Patients who have not recovered from > grade 1 (NCI CTCAE) prior adverse events from any cancer therapy, except for alopecia
* Pregnant or breastfeeding women
* Known hypersensitivity to any component of RO5458640 or previous severe hypersensitivity reactions to monoclonal antibody therapy
* History of active seizure disorder
* History of CNS or leptomeningeal metastases, except for clinically stable disease for at least 3 weeks prior to first study drug
* Cardiovascular illness: CVA or MI < 6 months prior to study, CHF > NYHA Class 2, QTcF >480 msec.
* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | approximately 2 years
Dose Limiting Toxicity (DLT) according to CTEP Common Terminology Criteria for Adverse Events Version 4.0 | approximately 2 years
Maximum Tolerated Dose (MTD) | approximately 2 years

SECONDARY OUTCOMES:
Pharmacokinetics: area under the concentration - time curve (AUC) on two administration schedules | approximately 2 years
Tumor response according to RECIST criteria | approximately 2 years
Antigenicity: Human anti-human antibody [HAHA] profile | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Canada (2):
  - Ottawa, Ontario
  - Toronto, Ontario
- København Ø, Denmark
- Amsterdam, Netherlands